CLINICAL TRIAL: NCT00342992
Title: Alpha-Tocopherol, Beta-Carotene Cancer Prevention Study (ATBC Study) Population
Brief Title: Alpha-Tocopherol, Beta-Carotene Cancer Prevention (ATBC) Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995012; OH95-C-N012
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stroke; Diabetes Mellitus; Heart Disease; Cancer
Keywords: Vitamin E; Micronutrients; Genetics; Smoking; Biomarkers
MeSH Terms: conditions — Stroke; Diabetes Mellitus; Heart Diseases; Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Male smokers in Southwestern Finland

SUMMARY:
The project is a passive follow-up of the Alpha-Tocopherol, Beta-Carotene Cancer Prevention (ATBC) Study cohort. Originally, this was a large, randomized, double-blind, placebo-controlled, 2x2 factorial primary prevention trial testing the effects of alpha-tocopherol and beta-carotene supplementation on cancer incidence and mortality. The study was conducted in Finland as a collaboration between the U.S. National Cancer Institute (NCI) and the National Public Health Institute of Finland. NCI has maintained passive surveillance of the cohort through Finnish national registries, including the cancer registry.

The primary purpose of the ATBC cohort follow-up is to use the existing risk factor data and biological specimens (i.e., serum, whole blood, DNA, red blood cells, and toenails) to test hypotheses relevant to cancer etiology, survival, early detection, and prevention. These data and biospecimens continue to provide an invaluable resource for the study of biochemical, nutritional, genetic, and molecular hypotheses. These analyses are made all the more informative and powerful by the addition of cases identified annually during the follow-up period, and the research benefits from a longer pre-diagnosis period (now over 30 years).

DETAILED DESCRIPTION:
The ATBC study was a randomized, double-blind, placebo-controlled, primary prevention trial to determine whether daily supplementation with a-tocopherol, beta-carotene, or both would reduce the incidence of lung or other cancers among male smokers. Between 1985 and 1988, 29,133 men ages 50 to 69 years, who smoked at least five cigarettes per day, were recruited from southwestern Finland. Participants were randomly assigned to receive either a-tocopherol as dl-a-tocopheryl acetate (50 mg/day), beta-carotene as all-trans-beta-carotene (20 mg/day), both supplements, or placebo capsules for 5-8 years (median 6.1 years) through April 30, 1993. Post-intervention follow-up has continued through the Finnish Cancer Registry and other national registries, and epidemiological analyses continue to be conducted.

ELIGIBILITY:
* INCLUSION CRITERIA:

Current smokers (five or more cigarettes per day at study entry) from Southwestern Finland.

EXCLUSION CRITERIA:

* Females
* Proven malignancy (except nonmelanoma skin cancer or cancer in situ)
* Severe angina pectoris
* Chronic renal insufficiency
* Cirrhosis of the liver
* Chronic alcoholism
* Anticoagulant therapy
* Use of supplements containing vitamin E greater than 20 mg/day, or vitaming A greater than 20,000 IU/day, or beta-carotene greater than 6 mg/day

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male smokers in Southwestern Finland
Sampling Method: Non-Probability Sample
Enrollment: 29133 (Actual)
Dates: Start 1995-03-03 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Cancer | Annually
  Annual linkage with Finnish Cancer Registry

SECONDARY OUTCOMES:
Causes of mortality | Anually

CONTACTS AND LOCATIONS:
Overall Officials: Demetrius A Albanes, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institute of Health and Welfare, Helsinki, Finland, Helsinki, Finland

REFERENCES:
- [Background] The alpha-tocopherol, beta-carotene lung cancer prevention study: design, methods, participant characteristics, and compliance. The ATBC Cancer Prevention Study Group. Ann Epidemiol. 1994 Jan;4(1):1-10. doi: 10.1016/1047-2797(94)90036-1. PMID 8205268
- [Background] Alpha-Tocopherol, Beta Carotene Cancer Prevention Study Group. The effect of vitamin E and beta carotene on the incidence of lung cancer and other cancers in male smokers. N Engl J Med. 1994 Apr 14;330(15):1029-35. doi: 10.1056/NEJM199404143301501. PMID 8127329
- [Background] Heinonen OP, Albanes D, Virtamo J, Taylor PR, Huttunen JK, Hartman AM, Haapakoski J, Malila N, Rautalahti M, Ripatti S, Maenpaa H, Teerenhovi L, Koss L, Virolainen M, Edwards BK. Prostate cancer and supplementation with alpha-tocopherol and beta-carotene: incidence and mortality in a controlled trial. J Natl Cancer Inst. 1998 Mar 18;90(6):440-6. doi: 10.1093/jnci/90.6.440. PMID 9521168
- [Derived] Huang J, Hodis HN, Weinstein SJ, Mack WJ, Sampson JN, Mondul AM, Albanes D. Serum Metabolomic Response to Low- and High-Dose Vitamin E Supplementation in Two Randomized Controlled Trials. Cancer Epidemiol Biomarkers Prev. 2020 Jul;29(7):1329-1334. doi: 10.1158/1055-9965.EPI-20-0187. Epub 2020 Apr 20. PMID 32312759
- [Derived] Hemila H. Vitamin E and Mortality in Male Smokers of the ATBC Study: Implications for Nutritional Recommendations. Front Nutr. 2020 Mar 31;7:36. doi: 10.3389/fnut.2020.00036. eCollection 2020. PMID 32296711
- [Derived] Hemila H. The effect of beta-carotene on the mortality of male smokers is modified by smoking and by vitamins C and E: evidence against a uniform effect of nutrient. J Nutr Sci. 2020 Mar 11;9:e11. doi: 10.1017/jns.2020.3. PMID 32215208
- [Derived] Lai GY, Wang JB, Weinstein SJ, Parisi D, Horst RL, McGlynn KA, Mannisto S, Albanes D, Freedman ND. Association of 25-Hydroxyvitamin D with Liver Cancer Incidence and Chronic Liver Disease Mortality in Finnish Male Smokers of the ATBC Study. Cancer Epidemiol Biomarkers Prev. 2018 Sep;27(9):1075-1082. doi: 10.1158/1055-9965.EPI-17-0877. Epub 2018 May 2. PMID 29720370
- [Derived] Playdon MC, Moore SC, Derkach A, Reedy J, Subar AF, Sampson JN, Albanes D, Gu F, Kontto J, Lassale C, Liao LM, Mannisto S, Mondul AM, Weinstein SJ, Irwin ML, Mayne ST, Stolzenberg-Solomon R. Identifying biomarkers of dietary patterns by using metabolomics. Am J Clin Nutr. 2017 Feb;105(2):450-465. doi: 10.3945/ajcn.116.144501. Epub 2016 Dec 28. PMID 28031192
- [Derived] Miranti EH, Freedman ND, Weinstein SJ, Abnet CC, Selhub J, Murphy G, Diaw L, Mannisto S, Taylor PR, Albanes D, Stolzenberg-Solomon RZ. Prospective study of serum cysteine and cysteinylglycine and cancer of the head and neck, esophagus, and stomach in a cohort of male smokers. Am J Clin Nutr. 2016 Sep;104(3):686-93. doi: 10.3945/ajcn.115.125799. Epub 2016 Aug 17. PMID 27534643
- [Derived] Lai GY, Weinstein SJ, Taylor PR, McGlynn KA, Virtamo J, Gail MH, Albanes D, Freedman ND. Effects of alpha-tocopherol and beta-carotene supplementation on liver cancer incidence and chronic liver disease mortality in the ATBC study. Br J Cancer. 2014 Dec 9;111(12):2220-3. doi: 10.1038/bjc.2014.514. Epub 2014 Oct 14. PMID 25314069
- [Derived] Moy KA, Mondul AM, Zhang H, Weinstein SJ, Wheeler W, Chung CC, Mannisto S, Yu K, Chanock SJ, Albanes D. Genome-wide association study of circulating vitamin D-binding protein. Am J Clin Nutr. 2014 Jun;99(6):1424-31. doi: 10.3945/ajcn.113.080309. Epub 2014 Apr 16. PMID 24740207
- [Derived] Mondul AM, Sampson JN, Moore SC, Weinstein SJ, Evans AM, Karoly ED, Virtamo J, Albanes D. Metabolomic profile of response to supplementation with beta-carotene in the Alpha-Tocopherol, Beta-Carotene Cancer Prevention Study. Am J Clin Nutr. 2013 Aug;98(2):488-93. doi: 10.3945/ajcn.113.062778. Epub 2013 Jun 26. PMID 23803886
- [Derived] Major JM, Yu K, Chung CC, Weinstein SJ, Yeager M, Wheeler W, Snyder K, Wright ME, Virtamo J, Chanock S, Albanes D. Genome-wide association study identifies three common variants associated with serologic response to vitamin E supplementation in men. J Nutr. 2012 May;142(5):866-71. doi: 10.3945/jn.111.156349. Epub 2012 Mar 21. PMID 22437554
- [Derived] Hemila H, Kaprio J. Subgroup analysis of large trials can guide further research: a case study of vitamin E and pneumonia. Clin Epidemiol. 2011 Feb 15;3:51-9. doi: 10.2147/CLEP.S16114. PMID 21386974
- [Derived] Hemila H, Kaprio J. Vitamin E may affect the life expectancy of men, depending on dietary vitamin C intake and smoking. Age Ageing. 2011 Mar;40(2):215-20. doi: 10.1093/ageing/afq178. Epub 2011 Jan 17. PMID 21242192
- [Derived] Mannisto S, Kontto J, Kataja-Tuomola M, Albanes D, Virtamo J. High processed meat consumption is a risk factor of type 2 diabetes in the Alpha-Tocopherol, Beta-Carotene Cancer Prevention study. Br J Nutr. 2010 Jun;103(12):1817-22. doi: 10.1017/S0007114510000073. Epub 2010 Feb 26. PMID 20187985
- [Derived] Hemila H, Kaprio J. Vitamin E supplementation and pneumonia risk in males who initiated smoking at an early age: effect modification by body weight and dietary vitamin C. Nutr J. 2008 Nov 19;7:33. doi: 10.1186/1475-2891-7-33. PMID 19019244
- [Derived] Kataja-Tuomola M, Sundell JR, Mannisto S, Virtanen MJ, Kontto J, Albanes D, Virtamo J. Effect of alpha-tocopherol and beta-carotene supplementation on the incidence of type 2 diabetes. Diabetologia. 2008 Jan;51(1):47-53. doi: 10.1007/s00125-007-0864-0. Epub 2007 Nov 10. PMID 17994292